CLINICAL TRIAL: NCT05849805
Title: The Feasibility, Safety and Efficacy of Y-3 Injection Through Skull Bone Marrow Bypassing Blood-brain Barrier in the Treatment of Acute Malignant Middle Cerebral Artery Infarction(SOLUTION)
Brief Title: Y-3 Injection Through Skull Bone Marrow in the Treatment of Acute Malignant Middle Cerebral Artery Infarction (SOLUTION)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, yilong Wang, Vice President of Beijing Tiantan Hospital, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY2023-052-02
Record Dates: First submitted 2023-04-06; First posted 2023-05-09 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Stroke, Acute Ischemic
Keywords: malignant middle cerebral artery infarction; Y-3; postsynaptic density protein 95 inhibitor; BBB-bypassing route; brain drug delivery; Intracalvaria bone marrow injection
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intracalvaria bone marrow injection group (Experimental): Y-3 ，Intracalvaria bone marrow injection , continuous medication for 3 days, with standard treatment and management according to the related guidelines.
  Interventions: Procedure: Intracalvaria bone marrow injection; Other: Conventional treatment
- Conventional treatment group (Sham Comparator): standard treatment and management according to related guidelines
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Procedure: Intracalvaria bone marrow injection — Intracalvaria bone marrow injection Y-3 (dose was given at 32 ug/kg), continuous medication for 3 days
  Arms: Intracalvaria bone marrow injection group
Other: Conventional treatment — standard treatment and management according to related guidelines

SUMMARY:
The mortality of malignant middle cerebral artery infarction (mMCAI) is up to 80%, while current available treatment is limited. The purpose of this study is to explore the feasibility, safety and efficacy of Intracalvaria bone marrow injection of cytoprotective drug Y-3 in mMCAI patients with contradictions of reperfusion therapy or poor reperfusion outcome.

DETAILED DESCRIPTION:
The mortality rate of malignant middle cerebral artery infarction (mMCAI) is up to 80%, while current available treatment is limited. Mainstream therapeutics include endovascular reperfusion therapy and decompressive craniectomy. But endovascular-reperfusion has limits such as short time window and hemorrhagic transformation risk, while decompressive craniectomy can reduce mortality but not infarct volume. Curative effect of intravenous injection of neuroprotective drugs is severely limited because of the blood-brain barrier. Microchannels connecting the skull bone marrow and dura may be effective drug delivery shortcuts bypassing the blood-brain barrier. Cytoprotective drug Y-3 affects dual aspects of ischemic cascade by disrupting both function of the synaptic folding post-synaptic density protein 95 (PSD-95), as well as α2-γ⁃Aminobutyric acid type A receptor （α2-GABAAR） agonist. Preclinical testing proved that intracalvaria bone marrow injection of Y-3 solution 24h post rat permanent middle cerebral artery infarction reduced rat infarction volume and improved neurological function.

The purpose of this study is to explore the feasibility, safety and efficacy of Intracalvaria bone marrow injection of cytoprotective drug Y-3 in mMCAI patients with contradictions of reperfusion therapy or poor reperfusion outcome.

This is a prospective, randomized, open-label, blinded endpoint (PROBE) clinical trial. The trial planned to enroll 20 patients with mMCAI, aged 18-85 years, within 24 hours of onset, with contradictions of reperfusion therapy or poor reperfusion outcome.

Patients will be randomly assigned to one of the following 2 groups at 1:1 ratio.

Intracalvaria bone marrow injection group: intracalvaria bone marrow injection Y-3 (dose was given as 32 ug/kg)once a day for 3 consecutive days, as well as standard treatment and management according to the related guidelines.

Conventional treatment group: standard treatment and management according to related guidelines

Face to face interviews will be made on baseline, 4±1 days after randomization, 7±2 days after randomization, 14±2 days after randomization or discharge day, and 90 days after randomization.

The primary outcomes include feasibility outcomes and safety outcomes. Feasibility Outcomes include the internal plate of skull was drilled throughly, drug leakage during injection, the patient refused to continue, failure for other reasons during 3 days'treatment. Safety Outcomes includes Infection events (skin infection, osteomyelitis, or intracranial infection), symptomatic and non-symptomatic intracranial hemorrhage, moderate to severe bleeding(defined by the GUSTO), hepatic insufficiency, renal insufficiency during the treatment, severe or extremely severe anaemia (hemoglobin <60g / L), mortality, incidence of other adverse events / serious adverse events reported. The secondary outcomes include change of the NIHSS scores from baseline to 14±2 days or at discharge, the NIHSS scores improved by 4 points from baseline at 7±2 days, the NIHSS limb score improved by 2 points from baseline at 7±2 days, change of core infarction volume from baseline to 7±2 days, change of Glasgow Coma Scale (GCS) scores from baseline values to 14±2 days or at discharge, the modified Rankin Scale（mRS） 0-3 points at 90±7 days, Rate of decompressive hemicraniectomy according to guidelines within 90±7 days, Rate of decompressive hemicraniectomy within 90±7 days, neurological intensive care unit (NICU) hospitalization days, cost of the NICU hospitalization

Safety indicators will be compared using the Fisher exact probability method. Primary effectiveness measures will be tested by the t-test or the Wilcoxon rank-sum test. Secondary effectiveness measures will use the Fisher exact probability method, where the comparison of neurofunction scale or daily living energy scale will be performed using non-parametric analysis. NICU hospitalization days and NICU hospitalization costs differences will be compared using the t-test or Wilcoxon rank-sum test. All statistics will be two-sided, P <0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1.18-75 years old; 2.No gender limitation; 3.Pre-stroke mRS score <2 4. Randomization can be finished within 24 hours of stroke onset (onset time is defined as last-seen-well time) 5. Ischemic stroke in the middle cerebral artery(MCA) territory meeting the following characteristics: A. 15<NIHSS≤30 B. Imaging within 6h of onset indicated the core area of infarction (rCBF<30% volume in CTP)>1/2 MCA territory or ASPECTS score≤6 6.If endovascular-reperfusion therapy is performed, the treatment is not effective with one of the following conditions: A. The NIHSS score decreased≤4 and the total score was still>15 B. The NIHSS score progressed immediately after the therapy and the total score≤30 7. Informed consent signed

Exclusion Criteria:

1. Concurrent with one of the other cerebrovascular diseases of the following conditions:

   A.Acute cerebral hemorrhage or subarachnoid hemorrhage B. Acute posterior circulation infarction C.Other types of TOAST classification such as intracranial artery dissection, vasculitis and moyamoya disease
2. Hemorrhagic transformation in the infarct area, over 30% of the infarct area, and significant occupancy effect
3. Bilateral pupil fixation / pupillary reflex disappeared
4. Decompressive craniectomy was planned before randomization
5. Resistant hypertension (systolic> 200mmHg or diastolic> 110mmHg) or hypotension (systolic <70mmHg or diastolic <50mmHg)
6. Abnormal blood glycemia before randomization (random venous blood glucose <2.8 mmol/L or> 23 mmol/L)
7. Severe hepatic or renal insufficiency (Note: severe hepatic insufficiency refers to the ALT> 3 times the upper limit of normal or the AST > 3 times the upper limit of normal; severe renal insufficiency means the creatinine value> 1.5 times the upper limit of normal or GFR <40 ml/min/1.73m2)
8. Severe cardiac insufficiency before randomization (compliance with New York College of Cardiology (NYHA) Cardiac Function Class III, IV)
9. Dual antiplatelet (aspirin plus clopidogrel or ticagrelor or cilostazol) within 24 hours or tirofiban within 4 hours
10. Combining with contraindications for intra-diplo administration, such as skull fracture, skull infection, subdural / external hematoma, subscalp hematoma, scalp skin or subcutaneous infection, etc
11. Bleeding tendency (including but not limited to): platelet count <100×109 / L; received heparin within nearly 24h, APTT ≥35s; oral warfarin, INR>1.7; new-oral-anticoagulant orally; with direct thrombin or factor Xa inhibitor; Combining with coagulopathy such as hemophilia
12. presence of severe or very severe anemia (hemoglobin <60g / L)
13. Combining with respiratory failure, and still difficult to correct after endotracheal intubation or tracheotomy, requiring ventilator treatment
14. Combining with severe CNS degenerative disease, such as AD, PD and severe dementia from various causes
15. Combining with other organic diseases, such as malignancy, the patient's life expectancy is less than 3 months
16. Allergy to any component of the therapeutic drug
17. Other neuroprotective agents without guideline recommendations and with unknown mechanism of the most important component were used within 24 hours of onset
18. Patients with pregnancy, lactation, or a possible pregnancy and a planned pregnancy
19. Unable to comply with the trial protocol or follow-up requirements
20. Other circumstances deemed unsuitable by investigator
21. Also participate in other interventional clinical trials

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2023-11-06 (Actual); Study Completion 2024-01-07 (Actual)

PRIMARY OUTCOMES:
Failed of drilling | during 3 days of treatment
  The rate of the internal plate of skull was drilled through
Number of drug-leakage events | during 3 days of treatment
  Number of drug-leakage events
Patients' tolerance of therapy | during 3 days of treatment
  The number of patient who refused to continue the treatment because of the intolerance
Failed for other reasons | during 3 days of treatment
  Number of failed for other reasons
Rate of participants with infection events | within 90±7 days after randomization
  Rate of participants with infection events (including skin infection, osteomyelitis of skull, or intracranial infection)
Rate of intracranial hemorrhage | within 90±7 days after randomization
  Rate of symptomatic and non-symptomatic intracranial hemorrhage
Rate of bleeding | within 90±7 days after randomization
  Rate of bleeding (moderate to severe bleeding, defined by the GUSTO)
Rate of hepatic insufficiency | within 90±7 days after randomization
  Rate of hepatic insufficiency: Posttreatment retest alanine aminotransferase(ALT) or aspartate transaminase(AST) value exceeds 3 times the upper normal limit
Rate of renal insufficiency | within 90±7 days after randomization
  Rate of renal insufficiency: glomerular filtration rate (GFR)<40 ml/min/1.73m2 during the treatment
Anaemia | within 90±7 days after randomization
  Severe or extremely severe anaemia (hemoglobin <60g / L)
Mortality | within 90±7 days after randomization
  Mortality
Adverse events / serious adverse events | within 90±7 days after randomization
  Incidence of other adverse events / serious adverse events reported

SECONDARY OUTCOMES:
Change of the NIHSS scores from baseline | 14±2 days after randomization or at discharge
  Change of the NIHSS scores from baseline to 14±2 days or at discharge. The National Institutes of Health Stroke Scale (NIHSS) is a standardized neurological examination score that is a valid and reliable measure of disability and recovery after acute stroke. Scores range from 0 to 42, with higher scores indicating increasing severity.
Patients with symptoms improvement | baseline，7±2 days after randomization
  The NIHSS scores improved by 4 points from baseline at 7±2 days
Patients with limbs' symptoms improvement | baseline，at 7±2 days after randomization
  The NIHSS limb score improved by 2 points from baseline at 7±2 days
Change of core infarction volume from baseline | baseline，7±2 days after randomization
  The core infarction volume is determined on CTP image with rCBF<30%
Change of GCS scores from baseline | baseline, 14±2 days after randomization or at discharge
  The GCS is a validated and reliable scale to evaluate level of consciousness in patients. The scale assesses 3 functions: Eye Opening, Verbal Response, and Motor Response. GCS scores range from 15 (best) to 3 (worst).
90 days Functional improvement | 90±7 days after randomization
  The modified Rankin Scale 0-3 points at 90±7 days
Rate of decompressive hemicraniectomy according to guidelines | 90±7 days after randomization
  Rate of decompressive hemicraniectomy according to guidelines within 90±7 days
Rate of decompressive hemicraniectomy | 90±7 days after randomization
  Rate of decompressive hemicraniectomy
Days of NICU hospitalization | From date of randomization until the date of discharge or date of death from any cause, assessed up to 1 month
  Days of NICU hospitalization
The cost of the NICU hospitalization | From date of randomization until the date of discharge or date of death from any cause, assessed up to 1 month
  The cost of the NICU hospitalization
Patients with symptoms improvement | baseline，14±2 days after randomization
  The NIHSS scores improved by 4 points from baseline at 14±2 days
Patients with limbs' symptoms improvement | baseline，at 14±2 days after randomization
  The NIHSS limb score improved by 2 points from baseline at 14±2 days

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wijdicks EF, Sheth KN, Carter BS, Greer DM, Kasner SE, Kimberly WT, Schwab S, Smith EE, Tamargo RJ, Wintermark M; American Heart Association Stroke Council. Recommendations for the management of cerebral and cerebellar infarction with swelling: a statement for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2014 Apr;45(4):1222-38. doi: 10.1161/01.str.0000441965.15164.d6. Epub 2014 Jan 30. PMID 24481970
- [Background] Treadwell SD, Thanvi B. Malignant middle cerebral artery (MCA) infarction: pathophysiology, diagnosis and management. Postgrad Med J. 2010 Apr;86(1014):235-42. doi: 10.1136/pgmj.2009.094292. PMID 20354047
- [Background] Berge E, Whiteley W, Audebert H, De Marchis GM, Fonseca AC, Padiglioni C, de la Ossa NP, Strbian D, Tsivgoulis G, Turc G. European Stroke Organisation (ESO) guidelines on intravenous thrombolysis for acute ischaemic stroke. Eur Stroke J. 2021 Mar;6(1):I-LXII. doi: 10.1177/2396987321989865. Epub 2021 Feb 19. PMID 33817340
- [Background] Jadhav AP, Desai SM, Jovin TG. Indications for Mechanical Thrombectomy for Acute Ischemic Stroke: Current Guidelines and Beyond. Neurology. 2021 Nov 16;97(20 Suppl 2):S126-S136. doi: 10.1212/WNL.0000000000012801. PMID 34785611
- [Background] Wu S, Wu B, Liu M, Chen Z, Wang W, Anderson CS, Sandercock P, Wang Y, Huang Y, Cui L, Pu C, Jia J, Zhang T, Liu X, Zhang S, Xie P, Fan D, Ji X, Wong KL, Wang L; China Stroke Study Collaboration. Stroke in China: advances and challenges in epidemiology, prevention, and management. Lancet Neurol. 2019 Apr;18(4):394-405. doi: 10.1016/S1474-4422(18)30500-3. PMID 30878104
- [Background] Powers WJ, Rabinstein AA, Ackerson T, Adeoye OM, Bambakidis NC, Becker K, Biller J, Brown M, Demaerschalk BM, Hoh B, Jauch EC, Kidwell CS, Leslie-Mazwi TM, Ovbiagele B, Scott PA, Sheth KN, Southerland AM, Summers DV, Tirschwell DL. Guidelines for the Early Management of Patients With Acute Ischemic Stroke: 2019 Update to the 2018 Guidelines for the Early Management of Acute Ischemic Stroke: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2019 Dec;50(12):e344-e418. doi: 10.1161/STR.0000000000000211. Epub 2019 Oct 30. PMID 31662037
- [Background] Vahedi K, Hofmeijer J, Juettler E, Vicaut E, George B, Algra A, Amelink GJ, Schmiedeck P, Schwab S, Rothwell PM, Bousser MG, van der Worp HB, Hacke W; DECIMAL, DESTINY, and HAMLET investigators. Early decompressive surgery in malignant infarction of the middle cerebral artery: a pooled analysis of three randomised controlled trials. Lancet Neurol. 2007 Mar;6(3):215-22. doi: 10.1016/S1474-4422(07)70036-4. PMID 17303527
- [Background] Kolias AG, Kirkpatrick PJ, Hutchinson PJ. Decompressive craniectomy: past, present and future. Nat Rev Neurol. 2013 Jul;9(7):405-15. doi: 10.1038/nrneurol.2013.106. Epub 2013 Jun 11. PMID 23752906
- [Background] Chamorro A, Dirnagl U, Urra X, Planas AM. Neuroprotection in acute stroke: targeting excitotoxicity, oxidative and nitrosative stress, and inflammation. Lancet Neurol. 2016 Jul;15(8):869-881. doi: 10.1016/S1474-4422(16)00114-9. Epub 2016 May 11. PMID 27180033
- [Background] Ugalde-Trivino L, Diaz-Guerra M. PSD-95: An Effective Target for Stroke Therapy Using Neuroprotective Peptides. Int J Mol Sci. 2021 Nov 22;22(22):12585. doi: 10.3390/ijms222212585. PMID 34830481
- [Background] Zhou L, Li F, Xu HB, Luo CX, Wu HY, Zhu MM, Lu W, Ji X, Zhou QG, Zhu DY. Treatment of cerebral ischemia by disrupting ischemia-induced interaction of nNOS with PSD-95. Nat Med. 2010 Dec;16(12):1439-43. doi: 10.1038/nm.2245. Epub 2010 Nov 21. PMID 21102461
- [Background] Hill MD, Goyal M, Menon BK, Nogueira RG, McTaggart RA, Demchuk AM, Poppe AY, Buck BH, Field TS, Dowlatshahi D, van Adel BA, Swartz RH, Shah RA, Sauvageau E, Zerna C, Ospel JM, Joshi M, Almekhlafi MA, Ryckborst KJ, Lowerison MW, Heard K, Garman D, Haussen D, Cutting SM, Coutts SB, Roy D, Rempel JL, Rohr AC, Iancu D, Sahlas DJ, Yu AYX, Devlin TG, Hanel RA, Puetz V, Silver FL, Campbell BCV, Chapot R, Teitelbaum J, Mandzia JL, Kleinig TJ, Turkel-Parrella D, Heck D, Kelly ME, Bharatha A, Bang OY, Jadhav A, Gupta R, Frei DF, Tarpley JW, McDougall CG, Holmin S, Rha JH, Puri AS, Camden MC, Thomalla G, Choe H, Phillips SJ, Schindler JL, Thornton J, Nagel S, Heo JH, Sohn SI, Psychogios MN, Budzik RF, Starkman S, Martin CO, Burns PA, Murphy S, Lopez GA, English J, Tymianski M; ESCAPE-NA1 Investigators. Efficacy and safety of nerinetide for the treatment of acute ischaemic stroke (ESCAPE-NA1): a multicentre, double-blind, randomised controlled trial. Lancet. 2020 Mar 14;395(10227):878-887. doi: 10.1016/S0140-6736(20)30258-0. Epub 2020 Feb 20. PMID 32087818
- [Background] Daneman R, Prat A. The blood-brain barrier. Cold Spring Harb Perspect Biol. 2015 Jan 5;7(1):a020412. doi: 10.1101/cshperspect.a020412. PMID 25561720
- [Background] Terstappen GC, Meyer AH, Bell RD, Zhang W. Strategies for delivering therapeutics across the blood-brain barrier. Nat Rev Drug Discov. 2021 May;20(5):362-383. doi: 10.1038/s41573-021-00139-y. Epub 2021 Mar 1. PMID 33649582
- [Background] Charabati M, Rabanel JM, Ramassamy C, Prat A. Overcoming the Brain Barriers: From Immune Cells to Nanoparticles. Trends Pharmacol Sci. 2020 Jan;41(1):42-54. doi: 10.1016/j.tips.2019.11.001. Epub 2019 Dec 12. PMID 31839374
- [Background] Xie J, Shen Z, Anraku Y, Kataoka K, Chen X. Nanomaterial-based blood-brain-barrier (BBB) crossing strategies. Biomaterials. 2019 Dec;224:119491. doi: 10.1016/j.biomaterials.2019.119491. Epub 2019 Sep 14. PMID 31546096
- [Background] Herisson F, Frodermann V, Courties G, Rohde D, Sun Y, Vandoorne K, Wojtkiewicz GR, Masson GS, Vinegoni C, Kim J, Kim DE, Weissleder R, Swirski FK, Moskowitz MA, Nahrendorf M. Direct vascular channels connect skull bone marrow and the brain surface enabling myeloid cell migration. Nat Neurosci. 2018 Sep;21(9):1209-1217. doi: 10.1038/s41593-018-0213-2. Epub 2018 Aug 27. PMID 30150661
- [Background] Brioschi S, Wang WL, Peng V, Wang M, Shchukina I, Greenberg ZJ, Bando JK, Jaeger N, Czepielewski RS, Swain A, Mogilenko DA, Beatty WL, Bayguinov P, Fitzpatrick JAJ, Schuettpelz LG, Fronick CC, Smirnov I, Kipnis J, Shapiro VS, Wu GF, Gilfillan S, Cella M, Artyomov MN, Kleinstein SH, Colonna M. Heterogeneity of meningeal B cells reveals a lymphopoietic niche at the CNS borders. Science. 2021 Jul 23;373(6553):eabf9277. doi: 10.1126/science.abf9277. Epub 2021 Jun 3. PMID 34083450
- [Background] Pulous FE, Cruz-Hernandez JC, Yang C, Kaya Zeta, Paccalet A, Wojtkiewicz G, Capen D, Brown D, Wu JW, Schloss MJ, Vinegoni C, Richter D, Yamazoe M, Hulsmans M, Momin N, Grune J, Rohde D, McAlpine CS, Panizzi P, Weissleder R, Kim DE, Swirski FK, Lin CP, Moskowitz MA, Nahrendorf M. Cerebrospinal fluid can exit into the skull bone marrow and instruct cranial hematopoiesis in mice with bacterial meningitis. Nat Neurosci. 2022 May;25(5):567-576. doi: 10.1038/s41593-022-01060-2. Epub 2022 May 2. PMID 35501382
- [Background] Mazzitelli JA, Smyth LCD, Cross KA, Dykstra T, Sun J, Du S, Mamuladze T, Smirnov I, Rustenhoven J, Kipnis J. Cerebrospinal fluid regulates skull bone marrow niches via direct access through dural channels. Nat Neurosci. 2022 May;25(5):555-560. doi: 10.1038/s41593-022-01029-1. Epub 2022 Mar 17. PMID 35301477